CLINICAL TRIAL: NCT00413205
Title: A Double-blind, Placebo-controlled Efficacy (as Assessed by Post-bronchodilator FEV1) and Safety Study of RAR Gamma in Subjects With Smoking-related, Moderate to Severe COPD With Emphysema Receiving Concurrent Optimised COPD Drug Therapy.
Brief Title: TESRA: (Treatment of Emphysema With a Gamma-Selective Retinoid Agonist)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB19751
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema | interventions — Retinoic Acid Receptor gamma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): po daily
  Interventions: Drug: Placebo
- RAR Gamma (Experimental): 5mg po daily
  Interventions: Drug: RAR Gamma

INTERVENTIONS:
Drug: Placebo — po daily
  Arms: Placebo
Drug: RAR Gamma — 5mg po daily
  Arms: RAR Gamma

SUMMARY:
This 2 arm study will investigate the efficacy, safety and tolerability of RAR Gamma versus placebo in ex-smokers with moderate or severe emphysema treated with optimal COPD therapy. Following optimization of COPD therapy (up to 6 weeks) patients will be randomized to receive either RAR Gamma (5mg) or placebo once daily using a 2:1 ratio (active:placebo), in addition to their standard therapy. Following the double-blind treatment period, patients will enter a 4-week follow-up period. The anticipated time on study period is 1-2 years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients of >44 years of age, with >10 pack-year smoking history;
* women not of child-bearing potential;
* ex-smokers (must have stopped smoking for >=12 months) with clinical diagnosis of emphysema;
* willing to be switched to optimal COPD therapy.

Exclusion Criteria:

* off oral steroids >28 days prior to enrollment;
* >2 exacerbations of pulmonary symptoms requiring outpatient treatment, or >1 exacerbation requiring hospitalization, within 12 months prior to screening;
* exposure to synthetic oral retinoids in past 12 months;
* history of allergy or sensitivity to retinoids.

Min Age: 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2007-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Post-bronchodilator FEVI | At intervals throughout study, and 2 and 6 months after cessation of study drug

SECONDARY OUTCOMES:
DLCo, lung densitometry, SGRQ, lung volume, walk test, time to first COPD exacerbation. | At intervals throughout study
AEs, SAEs, retinoid side effects, lab parameters. | Thoughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (55):
- United States (12):
  - Birmingham, Alabama
  - Los Angeles, California
  - San Diego, California
  - Torrance, California
  - Denver, Colorado
  - Chicago, Illinois
  - Detroit, Michigan
  - Omaha, Nebraska
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Spartanburg, South Carolina
  - Houston, Texas
- Bulgaria (3):
  - Pleven
  - Rousse
  - Sofia
- Czechia (4):
  - Brno
  - Karlovy Vary
  - Ostrava
  - Prague
- Hungary (6):
  - Balassagyarmat
  - Budapest
  - Nyíregyháza
  - Pécs
  - Szombathely
  - Törökbálint
- Reykjavik, Iceland
- Israel (6):
  - Ashkelon
  - Haifa
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Italy (4):
  - Modena, Emilia-Romagna
  - Genoa, Liguria
  - Pavia, Lombardy
  - Pisa, Tuscany
- Latvia (2):
  - Daugavpils
  - Riga
- Poland (5):
  - Bialystok
  - Katowice
  - Lodz
  - Poznan
  - Warsaw
- South Africa (8):
  - Bellville
  - Bloemfontein
  - Cape Town
  - Centurion
  - Durban
  - eManzimtoti
  - Johannesburg
  - Worcester
- Ukraine (2):
  - Donetsk
  - Kiev
- United Kingdom (2):
  - Coventry
  - Liverpool